CLINICAL TRIAL: NCT04723472
Title: An Open Randomized Controlled Study of Bismuth Quadruple Therapy With Cefuroxime as Rescue Therapy for Helicobacter Pylori Infection
Brief Title: Bismuth Quadruple Therapy With Cefuroxime for Helicobacter Pylori Eradication Treatment
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Want to modify the study further
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/041
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-01

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic bismuth quadruple treatment group (Active Comparator)
  Interventions: Drug: Classic bismuth quadruple treatment
- Cefuroxime containing bismuth quadruple treatment group (Experimental)
  Interventions: Drug: Cefuroxime containing bismuth quadruple treatment

INTERVENTIONS:
Drug: Cefuroxime containing bismuth quadruple treatment — Cefuroxime containing bismuth quadruple treatment:
  Rabeprazole 20mg bid po, Colloidal Bismuth Pectin 200mg bid po, Cefuroxime 500mg bid po, Metronidazole 400mg tid po Treatment duration is 14 days.
  Arms: Cefuroxime containing bismuth quadruple treatment group
Drug: Classic bismuth quadruple treatment — Classic bismuth quadruple treatment:
  Rabeprazole 20mg bid po, Colloidal Bismuth Pectin 200mg bid po, Tetracycline 500mg qid po, Metronidazole 400mg tid po Treatment duration is 14 days.
  Arms: Classic bismuth quadruple treatment group

SUMMARY:
To observe the efficacy of cefuroxime-containing bismuth quadruple regimen in the eradication treatment of Helicobacter pylori, and to evaluate whether it can be used as a remedial treatment for Helicobacter pylori after initial or repeated treatment failure.

DETAILED DESCRIPTION:
Introducing cefuroxime into the remedy treatment of Helicobacter pylori, on the one hand, the investigators will observe whether cefuroxime can replace tetracycline like amoxicillin, on the other hand, the investigators will observe whether it can reduce the rate of adverse effects caused by tetracycline and avoid the allergy of penicillin. If the experiment is successful, it will provide an effective and safe second-line treatment for the majority of patients with failed treatment of Helicobacter pylori.

ELIGIBILITY:
Inclusion Criteria:

* Employees, family members, and patients with positive C13 breath test in our hospital;
* Has received one or more previous Helicobacter pylori eradication therapy (no use of cefuroxime or tetracycline), and the result is still positive by C13 breath test;
* Willing to undergo gastroscopy and HP cultivation and identification;
* Age 18-70, gender unlimited;
* Willing to participate in and cooperate with the study, and willing to sign the informed consent.

Exclusion Criteria:

* Drugs that may affect the study results, such as PPI, H2 blockers, bismuth agents, antibiotics, etc. were taken in the 4 weeks before enrollment;
* Patients with gastrointestinal malignancy tumor;
* Patients with gastrinoma;
* After gastric or esophageal surgery;
* Suffers from serious diseases of the heart, lung, kidney, liver, blood, nervous system, endocrine system or mental system;
* Patients with contraindications or previous allergic reactions to the drugs used in this study;
* Pregnant or breastfeeding women;
* Patients with other medical conditions that may increase the treatment side effects;
* Those who cannot give informed consent;
* Has participated in other drug trials within 3 months;
* Not considered suitable for participants by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of success rates after 14 days of eradicate treatment with helicobacter pylori using a bismuth quadruple regimen containing cefuroxime and a classic bismuth quadruple regimen | The duration of treatment is 14 days. A C13 UBT will be performed 1 month after treatment.
  The comparison of eradication rate (0-100%), it is better to have a higher eradication rate.

SECONDARY OUTCOMES:
The Success rate of cefuroxime-containing bismuth quadruple regimen in the treatment of refractory Helicobacter pylori after 14 days | A C13 UBT will be performed 1 month after treatment.
  The eradication rate of new regimen in refractory Helicobacter pylori treatment (0-100%)
In vitro culture and drug sensitivity test of Helicobacter pylori were conducted to observe the drug resistance rate of Helicobacter pylori to cefuroxime, tetracycline and metronidazole. | before the treatment
  The drug resistance rate of Helicobacter pylori to cefuroxime, tetracycline and metronidazole（0-100%）
Adverse effect rate and safety of cefuroxime-containing bismuth quadruple regimen and classical bismuth quadruple regimen in patients with refractory Helicobacter pylori. | one month after treatment.
  questionnaire ; follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Meidong Xu, Study Director — ShanghaiDongfang Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Guildline in patient consent form